CLINICAL TRIAL: NCT05043831
Title: Direct Selective Laser Trabeculoplasty for Primary Open Angle Glaucoma and Ocular Hypertension in Ethnic Chinese Population The Zhuiguang Trial
Brief Title: Direct Selective Laser Trabeculoplasty in Ethnic Chinese Population The Zhuiguang Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study didnt start and will be re-designed
Sponsor: BelkinVision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: China-2021-01
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is not aware if subject is treated with SLT or DSLT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Selective Laser Trabeculoplasty (DSLT) (Experimental): Subjects will be treated with DSLT
  Interventions: Device: DSLT
- Selective Laser Trabeculoplasty (SLT) (Active Comparator): Subjects will be treated with SLT
  Interventions: Device: DSLT

INTERVENTIONS:
Device: DSLT — Direct-SLT is applied via the limbus to the trabecular meshwork
  Other Names: SLT

SUMMARY:
The objective of this study is to evaluate the effectiveness (Intra-Ocular Pressure lowering) and safety of Direct Selective Laser Trabeculoplasty (DSLT) in ethnic Chinese subjects with Primary Open Angle Glaucoma or Ocular Hypertension.

DETAILED DESCRIPTION:
Glaucoma, which is very common disease in China, can result in blindness if left untreated and as such it is extremely important to diagnose and treat the condition.

Usually doctors treat the first symptoms of glaucoma or ocular hypertension by prescribing eye drops. Unfortunately, there can be side effects associated with the use of these eye drops and there are reports of non-compliance due to difficulties in inserting these drops, all of which can impact on how effective this treatment regimen is.

The purpose of this study is to assess how well the new automated DSLT device for laser treatment of glaucoma or ocular hypertension works in comparison with the standard SLT in ethnic Chinese population and determine that it is as effective in reducing intraocular pressure.

DSLT or SLT will be performed in the study eye according to the randomization assignment. Eligible patients who sign the informed consent will be enrolled at each of the study sites, and undergo a washout (in the case of being medicated). After washout there will be a baseline visit, where continued eligibility is confirmed. Following confirmation of continued eligibility, 50% of patients being randomized to each treatment group. Randomization will be to a pre-determined randomization list.

Only one eye per participant will be included in the study and they will be treated using either DSLT or SLT as per the randomized treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older, any gender, of Chinese Han ethnicity, with corrected visual acuity > 6/60 in both eyes
2. Open angle glaucoma including exfoliative or pigmentary glaucoma or ocular hypertension.
3. IOP ≥ 22mmHg to ≤35mmHg (after washout of any IOP-lowering medications) for participants.
4. Gonioscopically visible scleral spur for 360 degrees without indentation
5. Ability to visualize the peri-limbal sclera for 360 degrees (using a lid speculum)
6. Willing and able to participate in the 12-month study, to comply with the study procedures and to adhere to the follow-up schedule.
7. Participant capable of giving informed consent

Exclusion Criteria:

1. Contraindications to conventional laser trabeculoplasty (e.g., corneal abnormalities, etc.)
2. Angle Closure Glaucoma
3. Congenital or developmental glaucoma
4. Secondary glaucoma except exfoliative or pigmentary glaucoma
5. Presence of any Peripheral Anterior Synechiae (PAS) in the study eye
6. Inability to conduct a reliable visual field (defined as fixation losses, false positives or false negatives greater than 33%)
7. Any of the following visual field findings using the Humphrey visual field analyzer the SITA-standard 24-2 program:

   1. A visual field MD of worse than -12dB
   2. Greater than or equal to 75% of points depressed below the 5% level and greater than or equal to 50% of points depressed below the 1% level on the PD plot.
   3. At least 50% of points (i.e 2 or more) within the central 5 degrees with a sensitivity ≤0dB on the decibel plot
   4. Points within the central 5 degrees of fixation with a sensitivity <15 dB in both hemifields on the decibel plot
8. A visual field MD of worse than -12dB in the fellow eye
9. Cup:Disc Ratio of more than 0.8
10. More than three hypotensive medications required (combination drops are considered as 2 medications)
11. Prior incisional or laser glaucoma surgery (including previous SLT or LPI) in the study eye.
12. Prior corneal refractive surgery
13. Complicated cataract surgery ≤ 6 months prior to enrollment
14. Presence of visually significant cataract in the opinion of the investigator
15. Clinically significant disease in either eye as determined by the Investigator.
16. Clinically significant amblyopia in either eye
17. Dense pigmentation or haemorrhage in the peri-limbal conjunctiva or anterior sclera
18. Women who are pregnant or may become pregnant during the course of the study.
19. In the opinion of the investigator the participant might require other ocular surgery within the 12-month follow-up period, unless for further reduction of their IOP
20. Concurrent treatment with topical, nasal, inhaled or systemic steroids.
21. Uncontrolled systemic disease that could impact the ability of the participant to attend follow up visits as per the discretion of the investigator.
22. Participation in another clinical study, not including a GLAUrious sub-study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
IOP reduction from baseline to 6 months | 6 months
  The primary effectiveness endpoint is the difference between the two treatment groups' change-from-baseline IOP, where change-from-baseline is defined as the difference between baseline (washed out for medicated patients) IOP and (washed out for medicated patients) IOP measured at 6 months for each subject.

SECONDARY OUTCOMES:
Mean percentage IOP reduction | 3, 6, 12 months
  Mean percentage reduction in IOP at 3, 6 and 12 months.
Subjects with at least 20% IOP reduction | 6 months
  Proportion of subjects with at least 20% reduction in IOP from baseline
Change in medications | 12 months
  Number of glaucoma medications at 12 months as compared to screening/visit 1 (before treatment) and compared between groups.
Treatment failures | r months
  Proportion of subjects in each group who are treatment failures (either had an incisional glaucoma surgery during the 6 months follow-up period, or are treated at the 6 months visit with hypotensive drugs in an equal or higher number than in the screening visit).
Adverse events | 6, 12 months
  Proportion of ocular adverse events between the 2 arms at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sun Xinghuai, Prof., Principal Investigator — Fundan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Study did not enrol